CLINICAL TRIAL: NCT01404884
Title: A Prospective Study To Evaluate The Safety And Effectiveness Of The SUPRACOR Presbyopic Treatment Algorithm For Myopia And Myopic Astigmatism Using LASIK
Brief Title: SUPRACOR for Myopia and Myopic Astigmatism
Acronym: SUPRACOR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1105
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Myopia; Myopic Astigmatism; Presbyopia
Keywords: myopia; astigmatism; presbyopia; SUPRACOR; multifocal
MeSH Terms: conditions — Myopia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SUPRACOR (Experimental): Treatment arm consisting of patients with history of myopia or myopic astigmatism who are also diagnosed with presbyopia.
  Interventions: Procedure: SUPRACOR

INTERVENTIONS:
Procedure: SUPRACOR — The developed software algorithm uses the subjective refraction of the eye to create a treatment for the distance vision correction. In addition to the treatment for the distance vision an additional central ablation component will be added to address the near vision.
  Other Names: PresbyLASIK

SUMMARY:
This clinical study has been planned to evaluate the safety and effectiveness of the SUPRACR presbyopic excimer laser treatment algorithm for myopic eyes developed for applying to the cornea of the human eye in a single center.

The developed software algorithm uses the subjective refraction of the eye to create a treatment for the distance vision correction. This part of the treatment does not show any difference to a regular aspheric LASIK treatment for myopic cases.

In addition to the treatment for the distance vision an additional central ablation component will be added to address the near vision.

The study design is applied as a single center unilateral eye safety and effectiveness study of the SUPRACOR presbyopic algorithm for myopia with a 3 months postoperative follow up.

DETAILED DESCRIPTION:
Presbyopia is an age-related progressive decrease in the ability to bring near objects to clear focus. It is attributed to changes in the accommodative apparatus in the visual system which includes the ciliary muscle and crystalline lens. Current Presbyopia management includes bifocal or multifocal corrections in spectacles or contact lenses that provide good focus over a range of object distances.

Current LASIK refractive surgery algorithms using Excimer laser are a safe, effective, and precise way to treat ametropia in eyes with regular corneas. The LASIK procedure uses a microkeratome to create a lamellar resection of the cornea at an intended depth ranging from 90 to 160 microns. The microkeratome is designed to maintain a "hinge" of tissue so that a flap of corneal epithelium and superficial stroma can be lifted to expose deeper stromal tissue while remaining attached to the cornea. The ablative energy of the excimer laser is then applied directly on the exposed corneal stroma to remove the required amount of tissue for a given refractive error. The amount of corneal tissue to be removed is determined by the magnitude of refractive correction and treatment area (optic zone). Once the laser ablation is completed, the flap is repositioned over the residual stromal bed.

The presbyopic treatment consists of a standard aspheric treatment for distance vision and the so called SUPRACOR addition to correct near vision.

The SUPRACOR addition provides a multifocal ablation with a central near addition with an aberration controlled transition zone towards the periphery, thereby allowing good focus over a range of object distances. This approach showed good near visual performance in hyperopic eyes (see also section 2.1).

The SUPRACOR presbyopic treatment algorithm subject to this study has been specifically developed to prospectively generate a treatment file for the Technolas 217z100 laser that will provide Presbyopia correction among eyes with primary myopia or myopic astigmatism (distance correction).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 45 years old and not older than 85 years
* Subjects must read, understand, and sign an Informed Consent Form (ICF).
* Subjects must be willing and able to return for scheduled follow up examinations through 3 months after surgery.
* Subjects must have up to -7.0 diopters (D) of absolute spherical myopia (not spherical equivalent), with up to -4.0 D of refractive astigmatism (NOT corneal astigmatism) by manifest subjective refraction. The spherical equivalent and must be no more than -9.0 D.
* Subjects must have presbyopia as determined by an age-related need for optical aid(> +1.50 D) for reading with their best distance correction.
* Subjects who have be screened successfully for acceptance of the SUPRACOR simulation
* Subjects who are contact lens wearers must have gas permeable (GP) lenses discontinued for at least 3 weeks and soft lenses discontinued for at least 1 week prior to the preoperative evaluation in the eye to be treated.
* High contrast, manifest, best spectacle-corrected logMAR distance visual acuity (VA) must be correctable to at least 0.0 (20/20 or 6/6) in both eyes.

Exclusion Criteria:

* Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns of remaining corneal thickness below the flap postoperatively.
* Subjects for whom the preoperative assessment of the ocular topography indicates that one or both eyes are not suitable candidates for treatment based upon the suggested computer-simulated treatment plan (e.G. Keratoconus).
* Subjects with anterior segment pathology, including dry eye syndrome and cataracts which in the Investigator's opinion, would interfere with best spectacle-corrected VA (BSCVA) or a successful treatment.
* Subjects who have undergone previous intraocular or corneal surgery of any kind, including any type of excimer laser surgery for either refractive or therapeutic purposes. Previous LASIK treatment and standard cataract surgery is not an exclusion criteria

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The percentage of treated eyes with a best corrected high contrast distance VA of 20/25 or better | 3 Months

SECONDARY OUTCOMES:
The percentage of treated eyes within +/- 1.00D of target refraction | 3 Months
The percentage of treated eyes within +/- 0.50D of target refraction | 3 Months
The percentage of treated eyes with an uncorrected high contrast near VA of 20/40 or better | 3 Months
Stability analysis: change of <1D MRSE between two consecutive post-op visits | 3 Months
Loss of more than 2 lines in BCVA for distance vision | 3 Months
The percentage of treated eyes with an induced subjective manifest refraction cylinder not within +/- 2.00D | 3 Months
Cumulative incidence of AEs | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Castanera, M.D., Principal Investigator — Instituto Oftalmologico Castanera
Locations (1):
- Instituto Oftalmologico Castanera, Barcelona, Spain

REFERENCES:
- [Background] de Ortueta D. Is peripheral presbyLASIK a center-distance technique? J Refract Surg. 2008 Jun;24(6):561; author reply 562. doi: 10.3928/1081597X-20080601-01. No abstract available. PMID 18581778
- [Background] Pinelli R, Ortiz D, Simonetto A, Bacchi C, Sala E, Alio JL. Correction of presbyopia in hyperopia with a center-distance, paracentral-near technique using the Technolas 217z platform. J Refract Surg. 2008 May;24(5):494-500. doi: 10.3928/1081597X-20080501-07. PMID 18494342
- [Result] Epstein RL, Gurgos MA. Presbyopia treatment by monocular peripheral presbyLASIK. J Refract Surg. 2009 Jun;25(6):516-23. doi: 10.3928/1081597X-20090512-05. PMID 19603619
- [Result] Alio JL, Amparo F, Ortiz D, Moreno L. Corneal multifocality with excimer laser for presbyopia correction. Curr Opin Ophthalmol. 2009 Jul;20(4):264-71. doi: 10.1097/icu.0b013e32832a7ded. PMID 19537363
- [Result] Pinelli R. More on peripheral PresbyLASIK as a center-distance technique. J Refract Surg. 2008 Sep;24(7):665. doi: 10.3928/1081597X-20080901-04. No abstract available. PMID 18811107
- [Result] Ortiz D, Alio JL, Illueca C, Mas D, Sala E, Perez J, Espinosa J. Optical analysis of presbyLASIK treatment by a light propagation algorithm. J Refract Surg. 2007 Jan;23(1):39-44. doi: 10.3928/1081-597X-20070101-07. PMID 17269242